CLINICAL TRIAL: NCT05921266
Title: Urolithin A Supplementation to Improve Endothelial and Cerebrovascular Function in Middle-aged Adults With Obesity
Brief Title: Urolithin A Supplementation in Middle-aged Adults With Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: UA15561
Record Dates: First submitted 2023-06-12; First posted 2023-06-27 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Obesity; Vascular Dementia; Cognitive Impairment
Keywords: Obesity; Urolithin A; Middle aged; Flow-mediated dilation; Endothelial function; fNIRS; Nitric oxide; Vascular contributions to cognitive impairment and dementia
MeSH Terms: conditions — Obesity; Dementia, Vascular; Cognitive Dysfunction; Dementia | interventions — 3,8-dihydroxy-6H-dibenzo(b,d)pyran-6-one

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Dietary Supplement: Urolithin A
- Control (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Urolithin A — Participants in the intervention group will receive 500 mg of urolithin A twice daily for 4 weeks (1,000 mg daily in total). The supplement will be administered in the form of softgels (4 softgels daily).
  Arms: Intervention
Other: Placebo — Participants in the control group will receive 0 mg of urolithin A twice daily for 4 weeks. The placebo will be administered in the form of inactive capsules (4 capsules daily).
  Arms: Control

SUMMARY:
The goal of this clinical trial is to learn about the effect of urolithin A, a dietary supplement, on blood flow in middle-aged adults with obesity. The main question it aims to answer is:

- Does urolithin A supplementation improve blood flow in large and small blood vessels in middle-aged adults with obesity?

Participants will be asked to:

* Take the dietary supplement daily for 4 weeks
* Attend two study visits to have their blood vessels checked, answer questionnaires, and give a sample of blood

Researchers will compare people who took the dietary supplement with others who took a placebo to see if the blood flow in the blood vessels improved.

DETAILED DESCRIPTION:
This study aims to measure the effect of urolithin A supplementation on endothelial function, cerebral blood flow regulation, and serum biomarkers of NO bioavailability and mitochondrial function in middle-aged adults with obesity. Briefly, 54 adults aged 40-64 years of age with a body mass index equal to or greater than 30 kg/m2 will be recruited to participate in a double-blind placebo-controlled parallel study for 4 weeks. Participants will be randomly assigned to intervention or control group. Those in the intervention group will consume 1,000 mg of urolithin A daily in the form of softgel capsules, whereas those in the control group will consume a placebo. Data collection will occur at baseline (day 0) and endpoint (day 28). The investigators will compare outcomes between control and intervention group. Researchers expect that urolithin A supplementation in middle-aged adults with obesity improves endothelial function and cerebral blood flow regulation, and that this improvement is accompanied by changes in biomarkers of NO bioavailability and mitochondrial function.

ELIGIBILITY:
Inclusion Criteria:

* Age: 40-64 years old, inclusive
* Obesity [BMI ≥30 kg/m2]
* Ability to read, write, and speak English
* Competence to provide written informed consent

Exclusion Criteria:

* Pregnant or breastfeeding women, or women who intend to become pregnant within the study period
* History of uncontrolled hypertension
* History of uncontrolled type 1 or type 2 diabetes mellitus
* Significant cardiac disease or chest pain in the last 6 months
* History of untreated depression or anxiety
* History of cognitive impairment
* History of uncontrolled significant GI disease (e.g., IBS, Crohn's disease)
* Allergy or intolerance to one or more of the intervention components
* Undergoing treatment for active cancer
* History of neurodegenerative disorders (e.g., multiple sclerosis)
* Presence of any condition affecting swallowing ability
* Any other medical condition that the investigators deem would adversely affect the participant's safety or ability to complete the study

Ages: 40 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2025-05-14 (Actual); Study Completion 2025-05-14 (Actual)

PRIMARY OUTCOMES:
Change in arterial function and local stiffness | Baseline (day 0) and endpoint (day 28)
  Flow-mediated dilation

SECONDARY OUTCOMES:
Change in blood flow on the surface of the hand | Baseline (day 0) and endpoint (day 28)
  Laser speckle contrast imaging
Change in reactive hyperemia index | Baseline (day 0) and endpoint (day 28)
  EndoPAT
Change in homeostatic cerebral blood flow | Baseline (day 0) and endpoint (day 28)
  Functional near-infrared spectroscopy
Change in plasma biomarkers of NO homeostasis | Baseline (day 0) and endpoint (day 28)
  Asymmetrical dimethylarginine
Change in plasma biomarkers of NO homeostasis | Baseline (day 0) and endpoint (day 28)
  Endothelin-1
Change in plasma biomarkers of NO homeostasis | Baseline (day 0) and endpoint (day 28)
  Bioactive nitrogen oxides
Change in plasma biomarkers of mitochondrial function | Baseline (day 0) and endpoint (day 28)
  Acylcarnitines

OTHER OUTCOMES:
Body weight | Baseline (day 0) and endpoint (day 28)
Body fat percentage | Baseline (day 0) and endpoint (day 28)
  Bioelectric impedance
Waist circumference | Baseline (day 0) and endpoint (day 28)

CONTACTS AND LOCATIONS:
Overall Officials: Andriy Yabluchanskiy, MD, PhD, Principal Investigator — University of Oklahoma Health Science Center
Locations (1):
- Translational GeroScience Laboratory - O'Donoghue Research Building, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF
Time Frame: Starting 6 months after publication
Access Criteria: By request upon PI approval